CLINICAL TRIAL: NCT04936373
Title: Pregnancy-related VTE; Quality of Patients' Lives
Brief Title: Quality of Life of Patients With Pregnancy Related VTE
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Assistant Professor, Jordan University Hospital
Other Study IDs: Deanship Academic Research-T
Record Dates: First submitted 2021-06-12; First posted 2021-06-23 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Health, Subjective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study of the quality of life and problems experienced by patients who developed pregnancy related VTE. It involves patients seen at JUH in 2012-2020. A questionnaire will be filled by those patients and any other patients in Jordan. It was translated to an Arabic form from EQ-5D, VEINES-QOL/SYM questionnaire and PEmb-QoL. The quality of their lives will be assessed and the problems encountered are going to be analyzed to try to find some solutions. This project is going to be a national research project with the efforts to try to find common platforms for those patients and nidus to establish a national support group.

DETAILED DESCRIPTION:
Retrospective study and analysis using a questionnaire which will be distributed to patients. The patients' data and contact details (phone numbers, whatsApp, email address…) will be collected from their clinical records at the JUH hospital. The period 2012-2020 will be covered. The questionnaire link is; file:///C:/Users/user/Downloads/QoL-post-VTE-during-pregnancy-5.pdf and file:///C:/Users/user/Downloads/arabic%20questionnaire%20last%201.pdf

ELIGIBILITY:
Inclusion Criteria:

* pregnancy related event
* confirmed diagnosis by an objective diagnostic tool (Duplex ultrasonography, CT pulmonary angiography, spiral CT scan or ventilation perfusion scan)
* consent (acceptance) to participate was obtained
* alive patients

Exclusion Criteria:

* death
* an objective diagnostic tool could not be found to confirm the diagnosis
* their event was not related to pregnancy
* refusal to participate

Ages: 18 Years to 49 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Patients were identified by searching the hospital database. Those who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
leg pain | 6 months
  limited mobility (difficulty walking, climbing stairs, bending, kneeling, squatting)
Breathlessness | 6 months
  daily activities at work, home or social activities
difficulties completing duties at work | 6 months
  Cut down the amount of time you spent on work or other activities , Accomplished less than you would like

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Al-Husban University Naser, Amman
  - The University of Jordan, Amman